CLINICAL TRIAL: NCT03302182
Title: An Open-label, Randomized Bioequivalence Study of Ritonavir Versus NORVIR in Healthy Chinese Subjects
Brief Title: Bioequivalence Study of Ritonavir Versus NORVIR in Healthy Chinese Subjects
Acronym: RTV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZYYY-LTNW-BE-2017-05-2
Record Dates: First submitted 2017-09-30; First posted 2017-10-05 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fasting group (Experimental): During the study session, healthy subjects will be administered a single dose of Ritonavir Tablet 100mg or NORVIR tablet 100mg under fasting condition.
  For group1:
  cycle 1:Ritonavir Tablet 100mg cycle 2:NORVIR tablet 100mg
  For group2:
  cycle 1:NORVIR tablet 100mg cycle 2:Ritonavir Tablet 100mg
  Interventions: Drug: Ritonavir for cycle1 and NORVIR for cycle 2; Drug: NORVIR for cycle 1 and Ritonavir for cycle 2
- Fed group (Experimental): During the study session, healthy subjects will be administered a single dose of Ritonavir Tablet 100mg or NORVIR tablet 100mg under fed condition.
  For group3:
  cycle 1:Ritonavir Tablet 100mg cycle 2:NORVIR tablet 100mg
  For group4:
  cycle 1:NORVIR tablet 100mg cycle 2:Ritonavir Tablet 100mg
  Interventions: Drug: Ritonavir for cycle1 and NORVIR for cycle 2; Drug: NORVIR for cycle 1 and Ritonavir for cycle 2

INTERVENTIONS:
Drug: Ritonavir for cycle1 and NORVIR for cycle 2 — During the study session, healthy subjects will be administered a single dose of Ritonavir Tablet 100mg in cycle 1 and NORVIR tablet 100mg in cycle 2 .
Drug: NORVIR for cycle 1 and Ritonavir for cycle 2 — During the study session, healthy subjects will be administered a single dose of NORVIR Tablet 100mg in cycle 1 and Ritonavir tablet 100mg in cycle 2 .

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and bioequivalence of Ritonavir tablet 100 mg versus NORVIR 100 mg tablet in healthy Chinese adult participants under fasting or fed condition.

DETAILED DESCRIPTION:
The study design is an Open-Label Randomized, Single-Dose, 2-way Crossover Bioequivalence Study with a washout period of 6 days. During each session, the subjects will be administered a single dose of 100mg Ritonavir (one Ritonavir Tablet 100mg or one NORVIR Tablet 100mg) under fasting or fed condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers of 18-45 years old.
2. Male (weight ≥50kg);Female (weight ≥45kg)
3. Body mass index (BMI) between 19~28 kg/m2;
4. In good health as determined by a physician/investigator based on medical history, vital signs, electrocardiogram (ECG), laboratory tests and physical examination findings at screening;
5. Female participant with negative result of HCG test and agrees to use adequate contraception from signing of informed consent form throughout the duration of the study and for 6 months after the last dose of study drug;
6. Male participant agrees to use adequate contraception and have no plan to donate sperm from signing of informed consent form throughout the duration of the study and for 6 months after the last dose of study drug;
7. Subject who totally understand the aim and progress of this clinical trial, make decision by his/her free will, and signed a consent form to follow the progress;
8. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.

Exclusion Criteria:

1. Subject who cannot tolerate venipuncture.
2. Allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator;
3. Subject who has past or present history of any serious diseases, including (but not limited to) digestive, cardiovascular, respiratory, urinary, musculoskeletal, endocrine, psychiatric or neurological, hematologic, immunological or metabolic disorders;
4. Abnormal results of physical examination (hematology, urine test,blood biochemistry etc.), vital signs, laboratory profile, a 12-lead electrocardiogram (ECG) or x-ray with clinical significance.
5. A positive result in hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, a syphilis test, or an human immunodeficiency virus (HIV) test;
6. Women who is during lactation, pregnancy or plan to have baby recently.
7. Women with positive result of HCG test.
8. Subject who refuse to use adequate contraception from signing of informed consent form throughout the duration of the study and for 6 months after the last dose of study drug;
9. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as alcohol consumption exceeding 14 units per week) within 6 months preceding this study or is unwilling to agree to abstain from alcohol and drugs throughout the study;
10. Heavy smokers (>5 cigarettes per day) within 6 months preceding this study or is unwilling to agree to abstain from smoking throughout the study;
11. Positive test results for alcohol or drug at Screening;
12. History of hospitalization or surgery within 3 months preceding this study.
13. Blood donation within the last 2 months (>= 400 ml), or have a plan to donate blood within 1 month after this study;
14. Intake of any other drug which might influence the results of the trial during two weeks previous to the start of the study.
15. Participation in another study with an investigational drug within the last 3 months preceding this study;
16. History of gastrointestinal surgery, vagotomy, enterotomy or other surgery that may influence gastrointestinal motility,PH or gastrointestinal absorption.
17. Intake of grapefruit or orange (or other food containing grapefruit or orange) 3 days previous to the start of the study. Intake of tea,coffee or other drink containing coffee more than 1L per day.
18. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive Ritonavir.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Cmax | 36 hours post-dose on Day 1,7
  Maximum Observed Plasma Concentration for ritonavir
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Tmax | 36 hours post-dose on Day 1,7
  Time to Reach the Maximum Plasma Concentration
AUC(0-inf) | Time Frame: 36 hours post-dose on Day 1,7
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for ritonavir
AUC(0-36h) | 36 hours post-dose on Day 1,7
  Area Under the Plasma Concentration-Time Curve From Time 0 to 36 hours Postdose for ritonavir

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No